CLINICAL TRIAL: NCT00863668
Title: Decay Kinetics of HIV With the Integrase Inhibitor Raltegravir
Brief Title: Raltegravir Activity In Lymphoid Tissues
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0901M57887
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infection; HIV Infections
Keywords: Infection; HIV 1; HIV; treatment naive
MeSH Terms: conditions — HIV Infections; Infections | interventions — efavirenz; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium; Integrase Inhibitors; Colonoscopy; Biopsy; Histocompatibility Testing; Transdermal Patch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efavirenz (Active Comparator)
  Interventions: Drug: Efavirenz + Tenofovir DF/Emtricitabine; Procedure: Colonoscopy with biopsies; Procedure: Inguinal Lymph Node Excision
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir + Tenofovir DF/Emtricitabine; Procedure: Colonoscopy with biopsies; Procedure: Inguinal Lymph Node Excision

INTERVENTIONS:
Drug: Efavirenz + Tenofovir DF/Emtricitabine — 600mg QD for 52 weeks + 300mg/200mg QD for 52 weeks
  Other Names: Sustiva; EFV; Tenofovir; Tenofovir Disoproxil Fumarate; TDF; Emtriva; FTC; Truvada; Atripla; Nucleoside Reverse Transcriptase Inhibitor; NRTI; Non-Nucleoside Reverse Transcriptase Inhibitor; NNRTI
  Arms: Efavirenz
Drug: Raltegravir + Tenofovir DF/Emtricitabine — 400mg BID for 52 weeks + 300mg/200mg QD for 52 weeks
  Other Names: Isentress; MK-0518; Tenofovir; Tenofovir Disoproxil Fumarate; TDF; Emtriva; FTC; Truvada; Integrase Inhibitor; Nucleoside Reverse Transcriptase Inhibitor; NRTI
  Arms: Raltegravir
Procedure: Colonoscopy with biopsies — Day 0, Day 2, Day 7, Day 14, Week 52
  Other Names: Colonoscopy; Biopsy; Secondary; Lymphatic; Tissue; Gastrointestinal; GALT; Peyers; Patch; Lamina; Propria
Procedure: Inguinal Lymph Node Excision — Day 0, Day 2, Day 7, Day 14, Week 52
  Other Names: Secondary; Lymphatic; Tissue; Inguinal; Lymph; Node; LN; Excision; Biopsy

SUMMARY:
The reduction with antiretroviral therapy (ART) of HIV RNA in blood, and HIV RNA in infected cells and in viruses associated with the follicular dendritic cell (FDC) network in lymphatic tissues, typically follows a two-phase pattern of decline. The half-life of the first-phase is about 1 day and that of the second phase is about 14 days, with comparable estimates for first-phase decay in SIV-infected rhesus macaques.

While substantial evidence supports the current view that first-phase decay reflects the death of activated CD4+ T cells infected before ART was begun, the sources of viral RNA in the second phase have not as yet been conclusively established. Possible sources of viral RNA that have been invoked in mathematical models, or for which there is experimental evidence, include longer-lived infected cells such as macrophages and resting CD4+ T cells, dissociation of virus from the FDC network, and productively infected CD4+ T cells that are not subject to clearance by host immune responses because of waning levels of HIV antigen.

Raltegravir (MK-0518) belongs to a new class of integrase inhibitors that potently suppress HIV and SIV replication, and reportedly markedly alters the second phase HIV decline in a way that challenges the current view that longer-lived infected cells are the source of virus in this phase. While mathematical modeling of decay of HIV RNA in blood was most consistent with 1) cells newly infected by long-lived cells, or 2) from activation of latently infected cells with full-length unintegrated HIV DNA as a source of second phase virus, we think the data are also quite consistent with the greater efficacy of integrase inhibitors in a particular cell type and/or anatomic site such as the gut.

In this protocol we will test the hypothesis that the rapid decrease in HIV replication associated with raltegravir is due to a more complete suppression of viral replication in lymphatic compartments such as lymph nodes and gastrointestinal lymphatic tissue. We will also investigate compartment-specific intracellular levels of raltegravir to potentially explain differences in changes in these compartments.

DETAILED DESCRIPTION:
The study will evaluate rates of HIV elimination in peripheral blood in comparison to secondary lymphatic tissues, including inguinal lymph nodes (LN) and gastrointestinal lymphatic tissues (GALT). HIV-infected patients who are antiretroviral therapy (ART) naive and fit criteria to initiate ART will be randomized to either Truvada (tenofovir/emtricitabine) + Sustiva (efavirenz - 600mg qDAY orally - standard of care) or Truvada + Isentress (raltegravir - 400mg BID orally).

Patients will have a blood draw, a colonoscopy with biopsies, and inguinal lymph node excision at days 0, 2, 7, 14, and week 52. Plasma HIV RNA and CD4+ T cell quantitation will be performed conventionally. HIV mRNA will be quantitated in LN and GALT using in-situ hybridization (ISH). Immunohistochemistry (IHC) will be performed to quantitate changes in CD4+ cell numbers over time in tissues from each respective ART regimen.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive (proven serologically at the time of screen, unless evidence for seroconversion)
* Evidence of recent (proven seroconversion within 4 months) or acute infection (HIV antibody negative, HIV RNA positive), or CD4 T Cells > 350 in peripheral blood and plasma viral load > 100,000 copies/ml
* Antiretroviral therapy naive (no prior history of antiretroviral therapy)
* Negative pregnancy test for eligible women of childbearing potential

Exclusion Criteria:

* Contraindication to surgical and endoscopic procedures (as judged by the principal investigator)
* Psychiatric or psychological illness that would make adherence to protocol procedures unlikely
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Rate of HIV mRNA Decline Measured in Peripheral Blood | 1 year
Rate of HIV mRNA Expression Decline Measured in Lymphatic Tissues | 1 year
CD4+ T Cell Number Increase in Peripheral Blood Over Time | 1 year
CD4+ T Cell Increase Quantified in Lymphatic Tissues Over Time | 1 year

SECONDARY OUTCOMES:
Intracellular concentrations of antiretroviral drugs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Schacker, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Division of Infectious Diseases, Minneapolis, Minnesota, United States